CLINICAL TRIAL: NCT02779374
Title: Autologous Bone Marrow Transplantation for Treatment of Premature Ovarian Insufficiency
Brief Title: Autologous Bone Marrow Transplantation for Premature Ovarian Insufficiency
Acronym: BMT-POI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammad Abdel-Rahman Mohammad Ahmed, Doctor, South Valley University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBGYN002
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Premature Ovarian Failure
Keywords: ovarian insufficiency Bone Marrow
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous bone marrow transplantation (Experimental): autologous bone marrow will be given by intravenous infusion. the intervention will be preceded by a period of 6 months of follow up the a period of 12 months follow up
  Interventions: Other: Autologous bone marrow transplantation

INTERVENTIONS:
Other: Autologous bone marrow transplantation — Bone marrow aspiration of 10 ml/kg is done from the posterior iliac crest. The sample is put in sterile container with appropriate amount of heparin then filtered to remove bone spicules, fat, and cellular debris. The filtered sample is injected unprocessed in a peripheral vein. The process is done once.

SUMMARY:
Currently, There is no treatment for Premature ovarian insufficiency (POI). Very small embryonic-like stem cells (VSELs) are found in the ovary. VSELs are able to regenerate the affected ovary. Stimulation was achieved by injection of mesenchymal stem cells that is supposed to secrete trophic factors.

Numerous studies in mice have proved the efficacy of bone marrow transplantation (BMT) in resuming the ovarian function after chemotherapy-induced ovarian insufficiency.

Allogeneic BMT raised the moral conflict about the origin of the newly developed oocytes. Several small studies examined the use of autologous BMT both in animal and in human. The results of these studies were promising. Intravenous injection is simpler and less invasive than ovarian injection as the later involves the use of laparoscopy. However, intravenous injection has not tested until now.

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI) has no curative treatment until now. It was noticed that some cases of POI to recover spontaneously. Furthermore, the concept of fixed prenatal pool of oogonia has been challenged and postnatal neo-oogenesis is currently proved.

Very small embryonic-like stem cells (VSELs) are found in the ovary. VSELs are stem cells that have noticed to survive chemotherapy induced gonadal insufficiency. Data from animal studies showed that stimulation of these stem cells result in regeneration of the affected ovary. Stimulation was achieved by injection of mesenchymal stem cells that is supposed to secrete trophic factors.

Numerous studies in mice have proved the efficacy of bone marrow transplantation (BMT) in resuming the ovarian function after chemotherapy-induced ovarian insufficiency. These studies have been followed by researches on human being. Human studies included the use of stem cells from different sites including BM, adipose tissue, and umbilical cord.

Allogeneic BMT raised the moral conflict about the origin of the newly developed oocytes. Although studies proved that these newly developed oocytes to be genetically traced to the recipient; some other studies showed that the newly developed oocytes originate from the donor BM. Several small studies examined the use of autologous BMT both in animal and in human. The results of these studies were promising. Use of autologous BMT also avoids the need for chemotherapy for conditioning and other related complications associated with allogeneic BMT. Human studies mostly used the ovarian injection of the BM. Intravenous injection is simpler and less invasive than ovarian injection as the later involves the use of laparoscopy. However, intravenous injection has not tested until now.

ELIGIBILITY:
Inclusion Criteria:

* Women with POI: For the purpose of the research women is considered to have POI if she is aged less than 40 years and has amenorrhea of at least 4 month with FSH level above 25 IU/L (repeated twice >4 weeks apart).

Exclusion Criteria:

* Abnormal karyotype
* Previous pelvic or abdominal radiotherapy
* Previous surgical management of ovarian pathology
* Chronic disease: renal, liver, cardiac, malignancy

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
menses | 6 months
  return of menses in a woman with previous ameneorrhea of at least 4 months before recruitment and during the 6 months of the pretest period

SECONDARY OUTCOMES:
Pregnancy | 12 months
  Occurrence of pregnancy during the period of 12 months of the post-test follow up
FSH | 12 months
  normalization of FSH (below 10 IU/L)
Antimullarian hormone (AMH) | 12 months
  normalization of AMH (above 0.9 ng/mL)
follicular activity | 12 months
  Growth of ovarian follicles to a size at least 18 mm in diameter
Endometrial thickness | 12 months
  Increase in endometrial thickness at least 8 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad AM Ahmed, MD, Principal Investigator — Egypt, Qena, South Valley University, faculty of Medicine
Locations (1):
- South Valley University, Qena Faculty of Medicine, Obstetrics and Gynecology Department, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santiquet N, Vallieres L, Pothier F, Sirard MA, Robert C, Richard F. Transplanted bone marrow cells do not provide new oocytes but rescue fertility in female mice following treatment with chemotherapeutic agents. Cell Reprogram. 2012 Apr;14(2):123-9. doi: 10.1089/cell.2011.0066. PMID 22471934
- [Background] Dan S, Haibo L, Hong L. Pathogenesis and stem cell therapy for premature ovarian failure. OA Stem Cells 2014 Feb 10;2(1):4.
- [Background] Hershlag A, Schuster MW. Return of fertility after autologous stem cell transplantation. Fertil Steril. 2002 Feb;77(2):419-21. doi: 10.1016/s0015-0282(01)02987-9. PMID 11821109
- [Background] Vassena R, Eguizabal C, Heindryckx B, Sermon K, Simon C, van Pelt AM, Veiga A, Zambelli F; ESHRE special interest group Stem Cells. Stem cells in reproductive medicine: ready for the patient? Hum Reprod. 2015 Sep;30(9):2014-21. doi: 10.1093/humrep/dev181. Epub 2015 Jul 22. PMID 26202914
- [Background] Edessy M, Hosni HN, Shady Y, Waf Y, Bakr S, Kamel M. Autologous stem cells therapy, the first baby of idiopathic premature ovarian failure. Acta Medica International. 2016;3(1):19-23.
- [Background] Lee HJ, Selesniemi K, Niikura Y, Niikura T, Klein R, Dombkowski DM, Tilly JL. Bone marrow transplantation generates immature oocytes and rescues long-term fertility in a preclinical mouse model of chemotherapy-induced premature ovarian failure. J Clin Oncol. 2007 Aug 1;25(22):3198-204. doi: 10.1200/JCO.2006.10.3028. PMID 17664466
- [Background] Hanna CB, Hennebold JD. Ovarian germline stem cells: an unlimited source of oocytes? Fertil Steril. 2014 Jan;101(1):20-30. doi: 10.1016/j.fertnstert.2013.11.009. PMID 24382341
- [Background] Bhartiya D, Anand S, Parte S. VSELs may obviate cryobanking of gonadal tissue in cancer patients for fertility preservation. J Ovarian Res. 2015 Nov 17;8:75. doi: 10.1186/s13048-015-0199-2. PMID 26576728
- [Background] Ghadami M, El-Demerdash E, Zhang D, Salama SA, Binhazim AA, Archibong AE, Chen X, Ballard BR, Sairam MR, Al-Hendy A. Bone marrow transplantation restores follicular maturation and steroid hormones production in a mouse model for primary ovarian failure. PLoS One. 2012;7(3):e32462. doi: 10.1371/journal.pone.0032462. Epub 2012 Mar 7. PMID 22412875